CLINICAL TRIAL: NCT06074705
Title: A Phase 1, Multicenter, First-in-human Study of DS-1471a In Subjects With Advanced Solid Tumors
Brief Title: A Study of DS-1471a In Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated by the sponsor due to a business decision.
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS1471-079; 2024-517984-21-00 (EU CTIS Number); jRCT2031230234 (Other: jRCT Number)
Record Dates: First submitted 2023-09-29; First posted 2023-10-10 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced Solid Tumor; DS-1471a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1, Dose Escalation Cohort 1: DS-1471a (Experimental): Participants with locally advanced or metastatic tumors will receive intravenous DS-1471a.
  Interventions: Drug: DS-1471a
- Part 1, Dose Escalation Cohort 2: DS-1471a (Experimental): Participants with locally advanced or metastatic tumors will receive intravenous DS-1471a.
  Interventions: Drug: DS-1471a
- Part 1, Dose Escalation Cohort 3: DS-1471a (Experimental): Participants with locally advanced or metastatic tumors will receive intravenous DS-1471a.
  Interventions: Drug: DS-1471a
- Part 1, Dose Escalation Cohort 4: DS-1471a (Experimental): Participants with locally advanced or metastatic tumors will receive intravenous DS-1471a.
  Interventions: Drug: DS-1471a
- Part 1, Dose Escalation Cohort 5: DS-1471a (Experimental): Participants with locally advanced or metastatic tumors will receive intravenous DS-1471a.
  Interventions: Drug: DS-1471a
- Part 1, Dose Escalation Cohort 6: DS-1471a (Experimental): Participants with locally advanced or metastatic tumors will receive intravenous DS-1471a.
  Interventions: Drug: DS-1471a
- Part 2, Dose Expansion (Tumor-specific Cohort 1): DS-1471a (Experimental): Participants will receive intravenous DS-1471a at the maximum tolerated dose and/or recommended dose for expansion as established in Part 1 Dose Escalation.
  Interventions: Drug: DS-1471a
- Part 2, Dose Expansion (Tumor-specific Cohort 2): DS-1471a (Experimental): Participants will receive intravenous DS-1471a at the maximum tolerated dose and/or recommended dose for expansion as established in Part 1 Dose Escalation.
  Interventions: Drug: DS-1471a
- Part 2, Dose Expansion (Tumor-specific Cohort 3): DS-1471a (Experimental): Participants will receive intravenous DS-1471a at the maximum tolerated dose and/or recommended dose for expansion as established in Part 1 Dose Escalation.
  Interventions: Drug: DS-1471a

INTERVENTIONS:
Drug: DS-1471a — Intravenous administration on Day 1 of each 28-day cycle

SUMMARY:
This first-in-human (FIH) study will assess the safety, preliminary efficacy, pharmacokinetics (PK), and immunogenicity of DS-1471a in participants with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
The objectives of this multinational, multicenter, open-label, 2-part, dose-escalation and dose-expansion, FIH study of participants with locally advanced or metastatic solid tumors are to evaluate the safety, maximum tolerated dose (MTD), recommended dose for expansion phase, preliminary efficacy, PK, and immunogenicity of DS-1471a.

ELIGIBILITY:
Key Inclusion Criteria:

The clinical site will screen for the full inclusion criteria per protocol.

* Sign and date the informed consent form (ICF)
* Adults ≥18 years at the time the ICF is signed
* Has a histologically or cytologically documented, locally advanced, metastatic, or unresectable solid tumor that is refractory to or intolerable with standard treatment, or for which no standard treatment is available
* Has at least 1 measurable lesion according to RECIST v1.1 1 on computed tomography (CT) or magnetic resonance imaging (MRI)
* Is willing and able to provide tumor tissue (newly obtained or archived)
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1
* Life expectancy ≥3 months
* Has a left ventricular ejection fraction (LVEF) ≥50% within 28 days prior to Cycle 1 Day 1
* Required baseline local laboratory data (within 7 days prior to Cycle 1 Day 1) as prespecified in the protocol
* A female participant of childbearing potential is eligible to participate if the following conditions are met:

  * Not pregnant as confirmed by highly sensitive pregnancy test within 7 days prior to study drug administration (Cycle 1 Day 1)
  * Agrees to adhere to a highly effective contraceptive method and agrees not to donate eggs or freeze/store eggs, during the intervention period, and for 7 months following the last dose of study drug
* A male participant is eligible to participate if he agrees to the following during the intervention period and for 4 months following the last dose of study drug:

  * Avoid donating sperm
  * Adhere to either abstinence or use of a condom during intercourse with a nonparticipant of childbearing potential PLUS partner use of an additional contraceptive method
* Is willing and able to comply with scheduled visits, study drug administration plan, laboratory tests, other study procedures, and study restrictions
* Patients with liver cirrhosis and liver cancer may be eligible to participate if they meet additional protocol specified criteria

Key Exclusion Criteria:

The clinical site will screen for the full exclusion criteria per protocol.

* Has an inadequate treatment washout period prior to start of study treatment (Cycle 1 Day 1) as prespecified in the protocol
* Has history of or current presence of untreated central nervous system (CNS) metastases
* Has a history of leptomeningeal carcinomatosis
* Has a history of (non-infectious) interstitial lung disease (ILD) other than radiation pneumonitis, currently has ILD, or when suspected ILD cannot be ruled out by imaging at screening
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses
* Has any of the following within the past 6 months: cerebrovascular accident, transient ischemic attack, arterial thromboembolic event, or pulmonary embolism
* Has uncontrolled or clinically significant cardiovascular disease
* Is requiring chronic steroid treatment (>10 mg daily prednisone equivalents)
* Has multiple primary malignancies, except adequately resected non-melanoma skin cancer, curatively treated in situ disease, superficial cancer in the gastrointestinal tract curatively resected by endoscopic surgery, or any other solid tumors curatively treated with no evidence of recurrent disease for ≥3 years
* Has unresolved toxicities from previous anticancer treatment
* Exposure to another investigational medical product within 4 weeks prior to Cycle 1 Day 1 or current participation in other therapeutic investigational procedures
* Has an active, known, or suspected autoimmune disease
* Has evidence of ongoing uncontrolled systemic bacterial, fungal, or viral infection.
* Has an active hepatitis or uncontrolled hepatitis B or C infection, except for participants with hepatitis B infection that is controlled by antiviral therapy
* For the Dose Escalation phase, has human immunodeficiency virus (HIV) infection. For the Dose Expansion phase, has active or uncontrolled HIV infection with exceptions per protocol.
* Has received a live, attenuated vaccine (messenger RNA [mRNA] and replication-deficient adenoviral vaccines are not considered live, attenuated vaccines) within 30 days prior to first exposure to study drug (Cycle 1 Day 1)
* Female who is pregnant or breastfeeding or intends to become pregnant during the study
* Has psychological, social, familial, or geographical factors that would prevent regular follow-up
* Has prior or ongoing clinically relevant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the investigator's opinion, could affect the safety of the subject; alter the absorption, distribution, metabolism, or excretion of the study drug; or confound the assessment of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose-limiting Toxicities Following Treatment With DS-1471a (Dose Escalation) | Cycle 1: Baseline up to Day 28 (each cycle is 28 days)
Number of Participants With Treatment-emergent Adverse Events Following Treatment With DS-1471a (Dose Escalation and Expansion) | Baseline up to 60 months

SECONDARY OUTCOMES:
Best Overall Response (BOR) As Assessed by the Investigator in Participants Following Treatment With DS-1471a (Dose Escalation and Expansion) | Baseline up to 60 months
  Best overall response (BOR) is recorded from the start of study drug until documented progressive disease (PD) or start of any anticancer treatment, whichever occurs first. Confirmation of complete response (CR) or partial response (PR) is required. As per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1, CR is defined as a disappearance of all target lesions, PR is defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD (at least a 20% increase in the sum of diameters of target lesions).
Time to Response (TTR) As Assessed by the Investigator in Participants Following Treatment With DS-1471a (Dose Escalation and Expansion) | Baseline up to 60 months
  Time to response (TTR) is defined as the time from the start of study drug to the date of the first documentation of response (CR or PR) as assessed by the investigator. As per RECIST v1.1, CR is defined as a disappearance of all target lesions and PR is defined as at least a 30% decrease in the sum of diameters of target lesions.
Duration of Response (DoR) As Assessed by the Investigator in Participants Following Treatment With DS-1471a (Dose Escalation and Expansion) | Baseline up to 60 months
  Duration of response (DoR) is defined as the time from first documentation of CR or PR to the date of the first documentation of PD as assessed by the investigator or to the date of death due to any cause, whichever occurs first. As per RECIST v1.1, CR is defined as a disappearance of all target lesions and PR is defined as at least a 30% decrease in the sum of diameters of target lesions.
Progression-free Survival (PFS) of Participants With Advanced Solid Tumors Following Treatment With DS-1471a (Dose Escalation and Expansion) | Baseline up to 60 months
  Progression-free survival (PFS) is defined as the time from the start date of study drug to the date of the first documentation of objective PD as assessed by the investigator or to the date of death due to any cause, whichever occurs first. As per RECIST v1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions.
Overall Survival (OS) of Participants With Advanced Solid Tumors Following Treatment With DS-1471a (Dose Escalation and Expansion) | Baseline up to 60 months
  Overall survival (OS) is defined as the time from the date of the start of study drug to the date of death due to any cause.
Objective Response Rate (ORR) of Participants With Advanced Solid Tumors Following Treatment With DS-1471a (Dose Expansion) | Baseline up to 60 months
  Confirmed objective response rate (ORR) is defined as the proportion of participants who have a confirmed BOR of CR or PR as assessed by the investigator. As per RECIST v1.1, CR is defined as a disappearance of all target lesions and PR is defined as at least a 30% decrease in the sum of diameters of target lesions.
Disease Control Rate (DCR) of Participants With Advanced Solid Tumors Following Treatment With DS-1471a (Dose Expansion) | Baseline up to 60 months
  Disease control rate (DCR) is defined as the proportion of participants who have a BOR of CR, PR, or SD as assessed by the investigator. As per RECIST v1.1, CR is defined as a disappearance of all target lesions, PR is defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD (at least a 20% increase in the sum of diameters of target lesions).
Pharmacokinetic Analysis Maximum Plasma Concentration (Cmax) of DS-1471a | Cycle 1 (Days 1, 2, 4, 8, 15, and 22), Cycle 2 (Day 1), Cycle 3 (Days 1, 2, 4, 8, 15, and 22), Cycles 4, 6, and 8 (Day 1), each cycle is 28 days
Pharmacokinetic Analysis Time to Reach Maximum Plasma Concentration (Tmax) of DS-1471a | Cycle 1 (Days 1, 2, 4, 8, 15, and 22), Cycle 2 (Day 1), Cycle 3 (Days 1, 2, 4, 8, 15, and 22), Cycles 4, 6, and 8 (Day 1), each cycle is 28 days
Pharmacokinetic Analysis Area Under the Plasma Concentration-Time Curve of DS-1471a | Cycle 1 (Days 1, 2, 4, 8, 15, and 22), Cycle 2 (Day 1), Cycle 3 (Days 1, 2, 4, 8, 15, and 22), Cycles 4, 6, and 8 (Day 1), each cycle is 28 days
  Area under the plasma concentration-time curve up to the last quantifiable time (AUClast), area under the plasma concentration-time curve from the time of dosing to 28 day (AUC28d), and area under the plasma concentration-time curve during dosing interval (AUCtau) will be assessed.
Pharmacokinetic Analysis Trough Plasma Concentration (Ctrough) of DS-1471a | Cycle 1 (Days 1, 2, 4, 8, 15, and 22), Cycle 2 (Day 1), Cycle 3 (Days 1, 2, 4, 8, 15, and 22), Cycles 4, 6, and 8 (Day 1), each cycle is 28 days
Percentage of Participants With Anti-Drug Antibodies Against DS-1471a | Cycle 1 (Days 1 and 8), Cycle 2 and 3 (Day 1), and Cycle 4 and every 2 cycles thereafter (Day 1), each cycle is 28 days
  Anti-drug antibodies (ADA) incidence is defined as the proportion of participants having treatment-emergent ADAs.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Florida Cancer Specialist, Sarasota, Florida
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Japan (3):
  - National Cancer Center Hospital East, Chiba
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/